CLINICAL TRIAL: NCT02098993
Title: Unfractionated Heparin in Acute Chest Syndrome: A Pilot Feasibility Randomized Controlled Trial of Unfractionated Heparin vs. Standard of Care in Acute Chest Syndrome
Brief Title: Feasibility Study of Unfractionated Heparin in Acute Chest Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment.
Sponsor: Craig Seaman (Other)
Collaborators: Vascular Medicine Institute (Unknown)
Responsible Party: Sponsor-Investigator, Craig Seaman, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACS13090197
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Acute Chest Syndrome; Sickle Cell Disease
Keywords: Sickle cell disease; Acute chest syndrome; Hemoglobinopathy; Hemolytic anemia; Heparin; Anticoagulant
MeSH Terms: conditions — Acute Chest Syndrome; Anemia, Sickle Cell; Hemoglobinopathies; Anemia, Hemolytic | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unfractionated heparin (Experimental): Subjects will be randomized within 24 hours of diagnosis to one of two treatment arms, Arm A, anticoagulation and standard of care, or Arm B, no anticoagulation and standard of care. Weight-adjusted UFH will be given at doses of 80 units per kilogram followed by 18 units per kilogram per hour intravenously for 7 days, or until discharge, if discharge is shorter than 7 days. UFH will be monitored by standard protocol to maintain the activated partial thromboplastin time in the therapeutic range per institutional guidelines.
  The experimental arm will receive standard of care, too, which will include the following: intravenous fluids, antibiotics, supplemental oxygen, incentive spirometry, pain management, red blood cell transfusions, and exchange transfusions.
  Interventions: Drug: Unfractionated heparin
- Standard of care (No Intervention): Standard care will include the following: intravenous fluids, antibiotics, supplemental oxygen, incentive spirometry, pain management, red blood cell transfusions, and exchange transfusions.

INTERVENTIONS:
Drug: Unfractionated heparin
  Arms: Unfractionated heparin

SUMMARY:
The purpose of this study is to determine the feasibility of performing a larger multicenter phase III trial to assess the effects of unfractionated heparin (UFH) in acute chest syndrome (ACS). Prespecified feasibility criteria consists of the ability to enroll potential study participants, which includes the timely notification of hospitalized patients with ACS, the capacity to consent eligible individuals, and the ability to appropriately randomize eligible patients within 24 hours of diagnosis. Additional feasibility objectives involve ensuring appropriate eligibility criteria, proper administration of the study drug, and the ability to completely and accurately collect clinical data of interest. The final aim of our pilot study is to provide preliminary data, with respect to treatment effect and variance, to allow sample size calculation in a larger trial given the lack of data available to help guide this process. The investigators hypothesize that the use of UFH in ACS will result in a decrease in the duration of hospitalization and improve other clinical outcomes, such as the duration of hypoxemia and duration of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ACS defined as a new pulmonary infiltrate involving at least one segment of the lung on a chest x-ray or chest CT scan with 2 or more of the following: chest pain, tachypnea, dyspnea, cough, hypoxemia, or body temperature greater than or equal to 38.0 degrees Celsius
* Hemoglobin electrophoresis confirming HbSS, SC, or B0 (historical records sufficient)
* Age greater than or equal to 18

Exclusion Criteria:

* Any absolute contraindication to heparin
* Platelet count less than 50 per microliter (current admission)
* Historical diagnosis of moyamoya disease as documented in medical records
* Historical diagnosis of proliferative retinopathy as documented in medical records
* Current participation in a chronic exchange transfusion program
* Underlying hypercoagulable disorder other than sickle cell disease
* Currently receiving therappeutic anticoagulation
* Currently receiving antiplatelet agents
* Currently receiving estrogen containing oral contraceptives
* Chest CT scan documented PE performed as standard of care prior to study enrollment (current admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Seaman, MD, Principal Investigator — University of Pittsburgh; Margaret Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburg Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Unfractionated Heparin: Subjects will be randomized within 24 hours of diagnosis to one of two treatment arms, Arm A, anticoagulation and standard of care, or Arm B, no anticoagulation and standard of care. Weight-adjusted UFH will be given at doses of 80 units per kilogram followed by 18 units per kilogram per hour intravenously for 7 days, or until discharge, if discharge is shorter than 7 days. UFH will be monitored by standard protocol to maintain the activated partial thromboplastin time in the therapeutic range per institutional guidelines.
  The experimental arm will receive standard of care, too, which will include the following: intravenous fluids, antibiotics, supplemental oxygen, incentive spirometry, pain management, red blood cell transfusions, and exchange transfusions.
  Unfractionated heparin
Period: Overall Study
Arm/Group | Unfractionated Heparin | Standard of Care
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unfractionated Heparin | Standard of Care | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.25 (3.77) | 32 (18.52) | 30.43 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Hospital Discharge
Description: Duration of hospitalization
Time Frame: Until hospital discharge
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
hours | 279.43 (267.98) | 127.31 (137.70)

2. Secondary Outcome: Duration of Hypoxemia Assessed by Arterial Oxygen Saturation
Description: Arterial oxygen saturation less than 90%
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
hours | 117.62 (60.52) | 51.49 (44.79)

3. Secondary Outcome: Duration of Fever Assessed by Body Temperature
Description: Body temperature greater than or equal to 38.0 degrees Celsius
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
hours | 24.90 (29.69) | 0 (0)

4. Secondary Outcome: Duration of Leukocytosis Assessed by White Blood Cell Count
Description: White blood cell count greater than 10,000 per liter
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
hours | 117.52 (60.52) | 53.11 (25.06)

5. Secondary Outcome: Duration of Moderate to Severe Pain Assessed by Visual Analog Scale for Pain
Description: Score of 4 or greater on the Visual Analog Scale for pain
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
hours | 88.68 (72.77) | 117.52 (60.52)

6. Secondary Outcome: Opioid Administration Per Participant
Description: Total dose of opioids per participant
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
mg | 3,446.75 (4,465.93) | 1,166.67 (1,112.61)

7. Secondary Outcome: Units of Red Blood Cells Administered
Description: Total number of units of red blood cells
Time Frame: 7 days
Measure: Number; unit: units
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
units | 5 | 4

8. Secondary Outcome: Percentage of Participants Transferred to Intensive Care Unit
Time Frame: 7 days
Measure: Number; unit: percent of participants
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
percent of participants | 0 | 33

9. Secondary Outcome: Percentage of Participants Requiring Mechanical Ventilation
Time Frame: 7 days
Measure: Number; unit: percent of participants
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
percent of participants | 0 | 0

10. Secondary Outcome: Percentage of Participants Experiencing Multiorgan Dysfunction Syndrome
Description: Acute development of 2 or more organs or organ systems unable to maintain homeostasis in a critically ill individual
Time Frame: 7 days
Measure: Number; unit: percent of participants
Arm/Group | Unfractionated Heparin | Standard of Care
Number analyzed (Participants) | 4 | 3
percent of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Unfractionated Heparin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unfractionated Heparin (N=4) | Standard of Care (N=3)
epistaxis (Blood and lymphatic system disorders) | 1 (2) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT02098993/Prot_SAP_000.pdf